CLINICAL TRIAL: NCT02645045
Title: Evaluation of Factors Affecting the Tear-film Lipid Layer Thickness
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2015-1009
Record Dates: First submitted 2015-12-28; First posted 2016-01-01 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2017-01

CONDITIONS: Dry Eye Syndrome
Keywords: Dry eye; Lipiview; Tear Lipid Layer; meibomian gland dysfunction
MeSH Terms: conditions — Dry Eye Syndromes; Meibomian Gland Dysfunction

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Dry eye: Patients with dry eye syndrome
- normal: Patients without dry eye

SUMMARY:
In this study, the investigators aim to determine the effects of age, sex, history of ocular surgery and contact lens use, and ocular surface and meibomian gland parameters on the lipid layer thickness (LLT) in normal subjects and patients with dry eye syndrome. Patients with dry eye syndrome and subjects with a healthy ocular surface will be enrolled. All participant will underwent LLT measurement with a LipiView interferometer, tear meniscus height measurement using optical coherence tomography, tear film break-up time (TBUT) determination, corneal and conjunctival staining, Schirmer's test, examination of the lid margins and meibomian glands, and assessment using the Ocular Surface Disease Index(OSDI) questionnaire.

ELIGIBILITY:
Inclusion Criteria:

1. age over 19 years old, Patients with dry eye syndrome and normal subjects

Exclusion Criteria:

1. patients less than 18 years of age and patients with histories of ocular surgery within 3 months; ocular injury; and ocular diseases such as ocular infection, allergy, and autoimmune disease; and patients with the use of a punctal plug or topical ocular medications other than artificial tears.
2. Patients who used artificial tears were instructed not to apply them for at least 12 hours 99 before the examinations

Ages: 19 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: age over 19 years old, Patients with dry eye syndrome and normal subjects
Sampling Method: Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2015-12-11 (Actual); Primary Completion 2016-02-10 (Actual); Study Completion 2016-02-10 (Actual)

PRIMARY OUTCOMES:
Tear Lipid Layer thickness measurement with a LipiView interferometer | 1 day

SECONDARY OUTCOMES:
tear meniscus height measurement using optical coherence tomography | 1 day
Corneal and conjunctival erosion grade(oxford score) | 1 day
tear film break-up time (TBUT) | 1 day
Schirmer's test (lacrimal secretion test) | 1 day
evaluation of the score of lid margins and meibomian glands | 1 day
Ocular Surface Disease Index(OSDI) questionnaire | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Ophthalmology, Yonsei Univeristy College of Medicine, Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
no plan to share IPD

REFERENCES:
- [Background] Hom MM, Martinson JR, Knapp LL, Paugh JR. Prevalence of Meibomian gland dysfunction. Optom Vis Sci. 1990 Sep;67(9):710-2. doi: 10.1097/00006324-199009000-00010. PMID 2234831
- [Background] Knop E, Knop N, Millar T, Obata H, Sullivan DA. The international workshop on meibomian gland dysfunction: report of the subcommittee on anatomy, physiology, and pathophysiology of the meibomian gland. Invest Ophthalmol Vis Sci. 2011 Mar 30;52(4):1938-78. doi: 10.1167/iovs.10-6997c. Print 2011 Mar. No abstract available. PMID 21450915
- [Background] Tomlinson A, Bron AJ, Korb DR, Amano S, Paugh JR, Pearce EI, Yee R, Yokoi N, Arita R, Dogru M. The international workshop on meibomian gland dysfunction: report of the diagnosis subcommittee. Invest Ophthalmol Vis Sci. 2011 Mar 30;52(4):2006-49. doi: 10.1167/iovs.10-6997f. Print 2011 Mar. No abstract available. PMID 21450918
- [Background] McCulley JP, Shine WE. The lipid layer of tears: dependent on meibomian gland function. Exp Eye Res. 2004 Mar;78(3):361-5. doi: 10.1016/s0014-4835(03)00203-3. PMID 15106913